CLINICAL TRIAL: NCT02800434
Title: Clinical Evaluation of Bilateral Hand Allograft: Pilot Study of 7 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-176
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Amputation
Keywords: allograft; hands; immunosuppression; fMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hand allograft (Experimental)
  Interventions: Procedure: hand allograft

INTERVENTIONS:
Procedure: hand allograft

SUMMARY:
The double amputation of the forearms is a rare handicap that seriously impacts the autonomy and the quality of life of patients, social and familial exclusion, and dependence on third parties for everyday activities.

The management of these patients is nearly exclusively through the use of prostheses. Certain patients refuse this solution, or remain penalized by the absence of sensation, the lack of precision in movements, and body image issues related to the amputation; the double graft of hands and forearms may, in this circumstance, be the only solution.

The objective of this pilot study was designed to evaluate the cerebral plasticity of patients who undergo bilateral hand allograph

ELIGIBILITY:
Inclusion Criteria:

* double amputated patients
* minimum of 3 months and maximum of 3 years interval between amputation and graft
* adult aged 20 to 40 years
* psychological maturity
* written informed consent

Exclusion Criteria:

* mono amputated patients
* previous history of malignant tumor in remission for less than 5 years,
* malignant tumor
* previous psychiatric history
* American Society of Anesthesiology (ASA) score >2
* New York Heart Association (NYHA) >1
* nenal insufficiency
* severe hypertension

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
fMRI for evaluation of brain plasticity after transplant | 1 year
  Evaluation of brain plasticity after transplant

SECONDARY OUTCOMES:
Rejection | Every 6 months following graft up to 5 years
Adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BADET, Principal Investigator — Hospices Civils de Lyon - Service d'Urologie et Chirurgie de la Transplantion
Locations (1):
- Service d'Urologie et Chirurgie de la Transplantion, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petruzzo P, Gazarian A, Kanitakis J, Parmentier H, Guigal V, Guillot M, Vial C, Dubernard JM, Morelon E, Badet L. Outcomes after bilateral hand allotransplantation: a risk/benefit ratio analysis. Ann Surg. 2015 Jan;261(1):213-20. doi: 10.1097/SLA.0000000000000627. PMID 24646555